CLINICAL TRIAL: NCT01102998
Title: Assessment of Sleep Complaints in Brain Tumor Survivors
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PBTSLP
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Brain Tumors
Keywords: Sleep complaints; Brain Tumor Survivors
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brain Tumor Survivors: Brain tumor survivors ages 8 to 18 years who are at least 5 years post diagnosis and at least 2 years post active therapy or observation and their parents/guardians will be approached to participate during clinic visits.

SUMMARY:
Survivors of pediatric brain tumors are noted to have increased rates of excessive daytime sleepiness. However, very little data are available regarding the specific sleep disturbances of pediatric brain tumor survivors. Children ages 8 to 18 years of age who are at least 5 years from diagnosis and at least 2 years post treatment or observation only for a brain tumor will be targeted to assess the prevalence of sleep complaints.

The study focuses on the following objectives:

* To estimate sleep disturbance in a cohort of pediatric brain tumor survivors.
* Estimate the rates of parent- and self-reported excessive daytime sleepiness in pediatric brain tumors
* Estimate the rates of parent-reported sleep-disordered breathing, including snoring and witnessed apneas, in pediatric brain tumor survivors
* Estimate the rates of parent- and self-reported behavioral sleep problems, including nocturnal enuresis, bedtime resistance, nighttime awakenings, nightmares, and fatigue in pediatric brain tumor survivors.

The Study focuses on the following secondary objectives:

* To describe bedtime patterns and sleep hygiene of pediatric brain tumor survivors.
* Estimate the typical parent- and self-reported weekday sleep duration of pediatric brain tumor survivors
* Estimate the typical parent- and self-reported weekend sleep duration of pediatric brain tumor survivors and if it differs from the weekday sleep duration
* Estimate the typical parent- and self-reported consistency of sleep hygiene in pediatric brain tumor survivors

DETAILED DESCRIPTION:
This non-therapeutic single arm study will characterize the prevalence and types of sleep complaints of pediatric brain tumor survivors. Brain tumor survivors ages 8 to 18 years who are at least 5 years post diagnosis and 2 years post active therapy and their parents/guardians will be approached to participate during clinic visits. If the patient and guardian agree to participate, they will be administered three questionnaires in the clinic during the patient's visit. From the medical record, the following variables will be utilized to characterize the subjects and estimate which groups are at greatest risk of sleep disturbances:

* Specific brain tumor diagnosis
* Location of tumor (cerebral hemispheres, parasellar region, posterior fossa, or spine)
* Age at diagnosis
* Obesity status
* Treatment modality (surgery, radiation therapy, and/or chemotherapy vs. observation only)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥8 to ≤ 18 years of age
* Brain tumor survivor
* ≥5 years post diagnosis
* ≥2 years post active cancer-directed therapy or observation only
* Parents speak and read English fluently
* Potential participant reads English fluently
* Potential participant/guardian willing to sign consent

Exclusion Criteria:

* Survivor of any cancer other than a brain tumor.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children ages 8 to 18 years of age who are patients at St Jude Children's Research Hospital and are at least 5 years from diagnosis and at least 2 years post treatment or observation only for a brain tumor were targeted to assess the prevalence of sleep complaints.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2010-04; Primary Completion 2012-09 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Sleep disturbance in a cohort of pediatric brain tumor survivors. | 2 years
  * Estimate the rates of parent- and self-reported excessive daytime sleepiness in pediatric brain tumors
  * Estimate the rates of parent-reported sleep-disordered breathing, including snoring and witnessed apneas, in pediatric brain tumor survivors
  * Estimate the rates of parent- and self-reported behavioral sleep problems, including nocturnal enuresis, bedtime resistance, nighttime awakenings, nightmares, and fatigue in pediatric brain tumor survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Crabtree, Ph.D, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St . Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org